CLINICAL TRIAL: NCT06077682
Title: Tropicamide Versus Cyclopentolate for Cycloplegic Refraction in Pediatric Patients With Esotropia: A Randomized Clinical Trial
Brief Title: Cycloplegic Refraction in Pediatric Patients With Esotropia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Islamic Hospital, Jordan (Other)
Collaborators: Jordan University of Science and Technology (Other); Yarmouk University (Other)
Responsible Party: Principal Investigator, Hashem Abu Serhan, Dr. Hashem Abu Serhan, Hamad Medical Corporation
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Cycloplegic Refraction & ET
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Cycloplegia; Refractive Errors; Esotropia; Vision Disorders
Keywords: Vision; refractive error; cycloplegic agent; cycloplegia; esotropia; tropicamide; cyclopentolate
MeSH Terms: conditions — Refractive Errors; Esotropia; Vision Disorders | interventions — Cyclopentolate; Tropicamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclopentolate arm (Active Comparator): To study the effect of cyclopentolate 1% for cycloplegic refractions in pediatric populations with ET:
  Firstly, we instilled an anesthetic drop into patients' eyes. Secondly, 2 drops of cyclopentolate 1% (cyclogel) 5 minutes apart were instilled. Autorefraction was taken at 60 minutes after first drop instillation. Primary outcome: spherical equivalent (SE) of cycloplegic refraction at 60 minutes.
  Interventions: Drug: Cyclopentolate
- Tropicamide arm (Active Comparator): To study the effect of tropicamide 1% for cycloplegic refractions in pediatric populations with ET:
  Firstly, we instilled an anesthetic drop into patients' eyes. Secondly, 2 drops of tropicamide 1% (mydriacil) 5 minutes apart were instilled. Autorefraction was taken at 30 minutes after first drop instillation. Primary outcome: spherical equivalent (SE) of cycloplegic refraction at 30 minutes.
  Interventions: Drug: Tropicamide

INTERVENTIONS:
Drug: Cyclopentolate — Well-known eye drop used for cycloplegic refraction among children.
  Other Names: Cyclogel
  Arms: Cyclopentolate arm
Drug: Tropicamide — Well-known eye drop used for cycloplegic refraction among children.
  Other Names: Mydriacil
  Arms: Tropicamide arm

SUMMARY:
The primary outcome of this study is to compare cyclopentolate 1% and tropicamide 1% for cycloplegic refractions in pediatric populations with esotropia. This will be a prospective double-blinded randomized clinical trial (RCT), multi-center, with randomized sequencing of cycloplegic agent; each patient received one agent at one visit, and the other agent in the next visit (2 different visits ≥ 1 week apart) within 3 months.

DETAILED DESCRIPTION:
Many studies have been conducted over the last few decades to assess the need for cycloplegia in assessing refractive errors. Plenty of research on pediatric populations has demonstrated that a lack of cycloplegia may contribute to an overestimation of myopia prevalence or substantial mistakes in estimating the prevalence of emmetropia and hyperopia. (1,2) The amount of refractive error varies by individual, as well as the type of cycloplegic refractive error. (3) As a result, there is no reliable method for adjusting non-cycloplegic refractions to approximate cycloplegic refractions. Consideration should be given to the type of cycloplegic agent to be used, preferred dosing, optimal methods of instillation, indications for use, and potential side effects. Despite the fact that the benefits of a cycloplegic examination are undeniable, there is still some confusion and various practice methods when it comes to cycloplegic exams. (4) Although atropine is the most potent cycloplegic agent currently available in clinical practice, its long duration of action (up to 12 days) and well-known side effects have shifted clinical practice toward cyclopentolate use. Cyclopentolate has been shown to provide effective cycloplegia, even in patients with moderate to severe hyperopia, with a relatively short duration of action (up to 24 hours) and fewer side effects. Thus, since its introduction in 1951, cyclopentolate has largely replaced atropine as the standard of care for pediatric cycloplegic examination. (4,5,6) Nevertheless, numerous adverse effects of cyclopentolate for children have been observed, including dry mouth and skin, tachycardia, fever, hallucinations, delirium, restlessness, seizures, ataxia, acute midbrain hemorrhage, and even death. (7,8,9) Many studies compared cyclopentolate to tropicamide for cycloplegia. (10, 11, 12) Tropicamide, unlike cyclopentolate, is a cycloplegic with a rapid onset and a short duration of action lasting up to 6 hours. In addition, fewer side effects have been reported when compared to cyclopentolate. (3,11) According to the literature, cyclopentolate may cause +0.175 to +0.39 D more hyperopia than tropicamide, which is clinically insignificant. (10,11,13) Furthermore, it has been discovered that there is a strong correlation between the time spent waiting to complete the exam and patient satisfaction levels, so reducing the waiting time clearly increases satisfaction levels. (14, 15) Esotropia is a convergent misalignment of the visual axes. Esotropia can be categorized in a variety of ways, usually based on age of onset or underlying causes: Infantile esotropia or acquired esotropia or accommodative esotropia, either normal accommodative convergence/accommodation (AC/A) ratio or high AC/A ratio or partially accommodative esotropia or Nonaccommodative esotropia, and Sensory esotropia. (16) Prevalence estimates of strabismus range from 0.8% to 6.8% in different populations. In the United States, esotropia and exotropia have similar prevalence rates, whereas in Ireland esotropia has been reported five times more frequently than exotropia, and in Australia esotropia has been reported to be twice as frequent as exotropia. (17) The prevalence of esotropia in children increases with age (e.g., higher prevalence at 4 to 6 years compared with 6 to 11 months), moderate anisometropia, and moderate amounts of hyperopia. (18) The potential benefits of treatment for esotropia include promoting binocular vision and improving visual function in each eye. (19) If binocularity is achieved, the number of surgical procedures over a lifetime and overall cost to society may be reduced. (20) Fusion and stereopsis are necessary for some careers and may be useful in sports such as baseball and activities such as needlepoint and watching 3D movies. (21) The appearance of crossed eyes may reduce employment opportunities because of stigma and bias. (22) In addition, binocular alignment is important for the development of a positive self-image and enhances social interactions by normalizing appearance as well as eye contact. (23) In one study, children aged 5 years and older expressed a negative feeling about dolls that had been altered to be esotropic or exotropic. (24) In another study, elementary school teachers rated personal characteristics of children with esotropia and exotropia more negatively than orthotropic children. (25) In a sample of children enrolled in the Multi-ethnic Pediatric Eye Disease Study, strabismus was associated with a decreased general health-related quality of life in preschool children, based on the parents' proxy reporting. (26) Adequate cycloplegia is necessary for accurate retinoscopy in children because of their increased accommodative tone compared with adults. The aim of this randomized clinical trial (RCT) is to explore the cycloplegic effect of tropicamide versus cyclopentolate in refracting pediatric subjects with esotropia.

ELIGIBILITY:
Inclusion Criteria:

Alignment: subjects with esotropia Age: 3-16 years Brown irides; grade 4 and 5 using iris color classification system developed by Seddon et al Duration: 2 different visits ≥ 1 week apart within 3 months

Exclusion Criteria:

Abnormal red reflex (e.g., media opacity) History of heart or neurological diseases History of developmental delay History of a previous allergy to cycloplegic agents Presence of syndromes (e.g., Down's syndrome) History of intraocular surgery

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Spherical equivalent (SE) mean difference between cyclopentolate and tropicamide | 3 months
  To study the SE of each drug and compare the mean difference between cyclopentolate and tropicamide To study the SE of each drug and compare the mean difference between cyclopentolate and tropicamide To study the SE of each drug and compare the mean difference between cyclopentolate and tropicamide To study the SE of each drug and compare the mean difference between cyclopentolate and tropicamide To study the SE mean difference between cyclopentolate and tropicamide

SECONDARY OUTCOMES:
Amplitude of accommodation | 3 months
  To measure the depth of cycloplegia mean difference between cyclopentolate and tropicamide

CONTACTS AND LOCATIONS:
Locations (2):
- Yarmouk University, Irbid, Jordan
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
The results will be shared with the researchers, and the data will be available upon request from the corresponding author.